CLINICAL TRIAL: NCT00033228
Title: A Phase I/II Pilot Study Of Intranodal Delivery Of A Plasmid DNA (Synchrovax SEM Vaccine) In Stage IV Melanoma Patients
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Chief Scientific Officer, Mannkind Coorporation
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069252; CTL-26-35
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): The first cohort of 6 patients received 500 ug of Synchrovax SEM plasmid DNA vaccine. All patients were to be monitored for dose limiting toxicities DLTs) for a minimum of 2 weeks after their second infusion of vaccine on Day 15 before allowing patients to enroll at the next dose group. The decision to progress to the next dose group was to be based on occurrence of DLTs observed in 1 or fewer (<33%) patients of a 6 patient cohort.
  Interventions: Biological: MKC1106-MT
- Cohort 2 (Experimental): The second cohort of 6 patients received 1000 ug of Synchrovax SEM plasmid DNA vaccine. All patients were to be monitored for dose limiting toxicities DLTs) for a minimum of 2 weeks after their second infusion of vaccine on Day 15 before allowing patients to enroll at the next dose group. The decision to progress to the next dose group was to be based on occurrence of DLTs observed in 1 or fewer (<33%) patients of a 6 patient cohort.
  Interventions: Biological: MKC1106-MT
- Cohort 3 (Experimental): The third cohort of 6 patients received 1500 ug of Synchrovax SEM plasmid DNA vaccine. The maximum tolerated dose (MTD) was to be determined by the observation of DLT at each dose group.
  Interventions: Biological: MKC1106-MT

INTERVENTIONS:
Biological: MKC1106-MT — Cancer Vaccine, Immunotherapy, 500 ug
  Arms: Cohort 1
Biological: MKC1106-MT — Cancer Vaccine, Immunotherapy, 1000 ug
  Arms: Cohort 2
Biological: MKC1106-MT — Cancer Vaccine, Immunotherapy, 1500 ug
  Arms: Cohort 3

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Infusing the vaccine directly into a lymph node may cause a stronger immune response and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of intranodal Synchrovax SEM plasmid DNA vaccine in patients with stage IV melanoma.
* Determine the safety and tolerability of this drug in these patients.
* Determine the immunological response, as measured by changes in frequency of T cells specific against vaccine-encoded epitopes before and after treatment, in patients treated with this drug.
* Determine the clinical response, as measured by lactic dehydrogenase levels and radiologic assessment of lesions, in patients treated with this drug.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive Synchrovax SEM plasmid DNA vaccine by continuous intranodal infusion on days 1-4. Treatment repeats every 14 days for up to 4 courses in the absence of unacceptable toxicity. Patients with evidence of stable or responding disease are eligible for 4 additional courses of treatment.

Cohorts of 6 patients receive escalating doses of Synchrovax SEM plasmid DNA vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 10 days after the last dose of study drug.

PROJECTED ACCRUAL: A total of 6-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma
* Must have tumor tissue available for determining antigen expression

  * At least 10% of tumor cells must stain positive for Melan-A/Mart-1 by immunohistochemistry
* HLA-A2 positive
* No brain metastases unless completely resected or without evidence of disease after treatment

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* WBC at least 3,000/mm3
* Platelet count at least 75,000/mm3
* Hemoglobin at least 9 g/dL

Hepatic:

* SGOT and SGPT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* Bilirubin no greater than 1.5 times ULN
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal:

* Creatinine no greater than 1.5 times ULN
* Urea no greater than 2.6 times ULN

Other:

* Not pregnant, nursing, or planning to become pregnant within 6 months of treatment completion
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No medical, sociological, or psychological impediments that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* At least 4 weeks since prior immunomodulatory drugs
* No other concurrent immunotherapy
* No concurrent immunomodulatory drugs

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since prior systemic corticosteroids
* No concurrent systemic corticosteroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 4 weeks since prior investigational drugs
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-01; Primary Completion 2003-03 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study was to evaluate the safety and tolerability of Synchrovax® pSEM Vaccine measured by the adverse event and severe adverse event profile.

SECONDARY OUTCOMES:
The secondary objective of the study was to determine the immunological response of patients as measured by tetramer assay and to assess clinical response by LDH levels and radiological assessment of lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Chair — Mannkind Corporation
Locations (5):
- United States (5):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Earle A. Chiles Research Institute at Providence Portland Medical Center, Portland, Oregon